CLINICAL TRIAL: NCT02840968
Title: Influence of Mediterranean Diet on Phase Angle in a Sample of Adult Population: Results of a Pilot Study
Brief Title: Adherence to Mediterranean Diet and Phase Angle
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Prof. Silvia Savastano, Researcher/Adjunct Professor, Federico II University
Other Study IDs: 239/11
Record Dates: First submitted 2016-07-12; First posted 2016-07-21 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Mediterranean Diet; Phase Angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In this cross-sectional observational study the investigators evaluated the association between the adherence to the MD and PhA in a sample of adult population, stratified according to categories of sex, age, and BMI.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian Subjects
* Healthy Subjects (defined as absence of a clinical condition that potentially influences fluid balance, ie, renal, endocrine, or myocardial disease, ascertained by participant questionnaire)

Exclusion Criteria:

* Hypocaloric diet in the last three months or specific nutritional regimens, including vegan or vegetarian diets,
* Vitamin/mineral or antioxidant supplementation,
* Clinical conditions that could influence fluid balance, including liver or renal failure, cancer, and acute or chronic inflammatory diseases, based on a complete medical examination and laboratory investigations,
* Occasional or current of use of drugs that could influence fluid balance, including non-steroidal anti-inflammatory drugs, hormone replacement therapy, diuretics weight-loss medications, anticonvulsivants and psychotropic agents, laxative use,
* Altered thyroid hormone function tests or thyroid hormone treatment,
* Alcohol abuse according to the Diagnostic and Statistical Manual of Mental Disorders (DSM)-V diagnostic criteria,
* Patients with implanted pacemakers or defibrillators because of the theoretical possibility of interference with the device activity due to the field of current induced by the impedance measurements,
* Subjects underweight with BMI<18.5,
* Subjects dropped out from the study since they refused to participate.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Recruitment strategies included attendance at the outpatient obesity clinics at the investigators Department or the outdoor hospital of the Campus Salute. The study is part of a large database started in 2010 to investigate the health status of the general population of Campania Region as analysed by the free consultation, visit, and diagnostics for people coming to the outdoor hospital held in different public squares of the investigators Region.
Sampling Method: Non-Probability Sample
Enrollment: 1464 (Actual)
Dates: Start 2010-01; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Adherence to Mediterranean Diet by Predimed Questionnaire | January 2010 - May 2016
Phase Angle by Bioimpedance Analysis | January 2010 - May 2016